CLINICAL TRIAL: NCT06735885
Title: Stanford-Matter Neuroscience High-Resolution fMRI Advanced Neurofeedback Feasibility Trial (fMRI Neurofeedback) Medical
Brief Title: fMRI Neurofeedback With Matter Neuroscience App
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Professor and Associate Chair of Psychiatry & Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 77871
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Depression Mild; Depression; Depression Moderate
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Arm 1A. No home training, no neurofeedback, no photos, no repeated scans, personal photos (No Intervention): No home training, no neurofeedback, no photos, no repeated scans, personal photos
- Arm 1B. No home training no neurofeedback, repeated scans (Experimental): No home training no neurofeedback, repeated scans
- Arm 2. No home training, neurofeedback, stock photos, repeated scans (Experimental): No home training, neurofeedback, stock photos, repeated scans
- Arm 3. No home training, neurofeedback, personal photos, repeated scans (Experimental): No home training, neurofeedback, personal photos, repeated scans
- Arm 4. Home training, no neurofeedback, stock photos, repeated scans (Experimental): Home training, no neurofeedback, stock photos, repeated scans
- Arm 5. Home training, neurofeedback, stock photos, repeated scans (Experimental): Home training, neurofeedback, stock photos, repeated scans
- Arm 6. Home training, no neurofeedback, personal photos, repeated scans (Experimental): Home training, no neurofeedback, personal photos, repeated scans
- Arm 7. Home training, neurofeedback, personal photos, repeated scans (Experimental): Home training, neurofeedback, personal photos, repeated scans

INTERVENTIONS:
Device: Matter Neuroscience App — An iPhone smartphone application
Other: Stock Photos — Stock Photos
Other: No Home Training — No Home Training
Device: Personal Photos — Personal Photos
Other: Home Training — Home Training

SUMMARY:
Study will utilize an app, Matter Neuroscience, designed to help users with depression understand positive emotions and the neurotransmitters that create them. We hope to learn the safety and efficacy of neurofeedback for treating depression and lay the groundwork for a pivotal clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, between the ages of 18 and 80 at the time of screening.
2. Primary diagnosis of nonpsychotic major depressive disorder (MDD) without a history of psychotic features.
3. Score on the MADRS scale between 15-25
4. Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questionnaires / follow instructions during fMRI. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
5. Must possess an iPhone with the latest iOS version compatible with the app, and be capable of using the study app with the phone.
6. 1-5 lifetime adequate antidepressant medication failures (ATHF).
7. The dose of the primary antidepressant medication (if applicable) must be stable for 4 weeks prior to baseline, and participants must agree to continue at this dose throughout the study period.
8. In good general health, as evidenced by medical history and determined by study physician
9. For women of reproductive potential: agree to the use of highly effective contraception during study participation.
10. Adequate visual acuity (with or without corrective lenses) to view study materials while in the MRI.
11. Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

1. 1. Contraindication to MRI (ferromagnetic metal in their body)
2. Severe claustrophobia
3. Women that are pregnant or breastfeeding or with a positive urine pregnancy test at participation, or who are planning to become pregnant during the study period.
4. Primary psychiatric condition other than MDD requiring treatment except stable comorbid anxiety disorder
5. History of or current psychotic disorder, schizophrenia, psychosis, bipolar disorder, or severe borderline personality disorder.
6. Diagnosis of intellectual disability, autism spectrum disorder, or other neurodevelopmental disorder.
7. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
8. Urine screening test positive for recent use of recreational drugs.
9. Considered at significant risk for suicide during the course of the study.
10. Recent (within 4 weeks of any clinical effect) or concurrent use of rapid acting antidepressant agent (i.e., a course of ECT or TMS). Excluding ketamine.
11. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma as determined by the PD.
12. Untreated or insufficiently treated endocrine or metabolic disorder.
13. Any other condition deemed by the PD to interfere with the study or increase risk to the participant
14. Alexithymia as determined by the Toronto Alexithymia Scale
15. Treatment with an investigational drug or other intervention within the study period.
16. Not currently in a major depressive episode as defined by the MINI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and efficacy of neurofeedback for treating depression through MADRS scale changes | Screening, Baseline, Immediate Post, One Month Post, Optional Three Month and Optional Six Month
  Determine the safety and efficacy of neurofeedback for treating depression through MADRS (Montgomery-Åsberg Depression Rating Scale) scale changes.
  The 9-item self-report version of the MADRS has an overall score range from 0-27, with higher scores corresponding to higher levels of depression.

SECONDARY OUTCOMES:
Measure fMRI Change | Baseline, Week 2, Week 4, Week 6, Immediate Post, Optional Three Month Post Scan
  Measure fMRI Change

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, MD, Principal Investigator — Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine
Locations (1):
- Stanford University Brain Stimulation Lab, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided